CLINICAL TRIAL: NCT07026838
Title: Advancing Family Wellbeing Through a Massive Open Online Intervention: The LightBEAM Program Protocol for Randomized Waitlist Control Trial
Brief Title: Advancing Family Wellbeing Through a Massive Open Online Intervention: The LightBEAM Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other); Children's Hospital Research Institute of Manitoba (Other); Manitoba Centre for Health Policy (Unknown); George & Fay Yee Centre for Healthcare Innovation (Unknown)
Responsible Party: Principal Investigator, Leslie E. Roos, Associate Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LightBEAM; 435-2023-0637 (Other Grant/Funding Number: Social Sciences and Humanities Research Council of Canada (SSHRC) Insight Grant)
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Depression, Anxiety; Anger; Parenting; Stress Psychological; Parent Child Relationship; Child Development
Keywords: parenting; mental health; anxiety; depression; psychoeducation; massive online open intervention
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress, Psychological; Psychological Well-Being | interventions — Mental Health

STUDY DESIGN:
Intervention Model Description: Using a two-arm clinical design, participants will be randomized in a 1:1 allocation to receive either the 12-week LightBEAM program or the waitlist control. Co-parents will be assigned to the same condition as the parent participant who invited them to join the study. After the 12-week LightBEAM program has been completed by the intervention condition, participants in the waitlist control group will complete rthe baseline questionnaires again prior to gaining access to the LightBEAM intervention. Longitudinal self-report questionnaires will be administered digitally at three timepoints: pre-intervention, post-intervention and at six months follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The LightBEAM Program Group (Experimental): Participants will complete 12 weeks of the LightBEAM program. Participants will be instructed to move through the weekly videos and practice exercises at a self-guided pace. Each week of LightBEAM includes: (a) 12-16 minutes of therapeutic mental health and parenting video content, (b) exercises to practice key skills, (c) access to the online forum to cultivate social support through interaction with other parents and peer coaches, and (d) a brief in-app survey for progress monitoring.
  Interventions: Behavioral: The Light Building Emotional Awareness and Mental Health (BEAM) Program
- Waitlist Control Group (No Intervention): Participants in the waitlist control group will be informed via email that they have been assigned to the waitlist condition. Along with this notification, they will receive a list of Canada-wide mental health and parenting resources, which they may choose to access at their discretion. Participants will be instructed to continue with any existing services or support they are utilizing as usual during the wait period. Following the completion of the wait period, participants will be notified and provided access to begin the 12-week LightBEAM program. Once enrolled in LightBEAM participants will complete 12 weeks of the LightBEAM program.

INTERVENTIONS:
Behavioral: The Light Building Emotional Awareness and Mental Health (BEAM) Program — The LightBEAM Program builds on mHealth best practices and evidence-based program design principles with the core objectives of improving parental mental health and fostering supportive parenting. Program content draws on transdiagnostic emotion-focused mental health and third wave Cognitive Behavioural Therapy principles such as Dialectical Behavioural Therapy, Acceptance and Commitment Therapy.
  Program delivery will be facilitated through a mobile application. The LightBEAM program consists of four different components; weekly parenting and mental health videos, weekly progress tracking, a group forum, and exercises designed to reinforce skills learned through the video content.
  Arms: The LightBEAM Program Group

SUMMARY:
Early childhood is a critical period for developmental outcomes, and the parent-child relationship plays a vital role in shaping cognitive and social development. However, elevated parental distress (e.g., depression, anxiety, anger) can disrupt healthy relationships, increasing the risk of negative child outcomes such as difficult temperaments, altered cognitive development, and socio-emotional challenges. Despite the well-documented effects of untreated parental distress, Canadian families face significant barriers to accessing timely and effective mental health support. To address this gap, our team developed BEAM, an app-based program that provides parenting and mental health resources. BEAM includes expert-led videos, online forums, progress monitoring, and peer-coaching sessions. Clinical trials to date evaluating BEAM have shown promising results, demonstrating reductions in parent depression, anxiety, and harsh parenting practices. Building on BEAM's success, we have developed the LightBEAM program, which aims to expand these supports into a scalable, accessible, massive online open intervention (MOOI) to reach a larger number of families across Canada, particularly in underserved areas or those on waitlists for individualized services. LightBEAM has the potential to support parental mental health, fostering healthier child and family development while addressing barriers to traditional mental health care. This trial involves a pre-post randomized trial design with primary aims of (1) assessing feasibility and acceptability metrics of LightBEAM including recruitment/retention, sustainability, satisfaction, and unmet needs, (2) examining the efficacy of LightBEAM versus waitlist control at improving family and mental health outcomes, and (3) determine for whom LightBEAM is more or less effective at engaging with and addressing mental health needs.

This trial will evaluate the feasibility and effectiveness of LightBEAM with a sample of up to 300 parent participants with a child aged 18-107 months. Co-parents of parent participants are permitted to participate in the study as well but are not included in this sample of 300 parent participants. Study participants will complete 12 weeks of psychoeducation modules in the BEAM app. The LightBEAM program will consist of four different components; weekly parenting and mental health videos, weekly progress tracking, a group forum, and exercises designed to reinforce skills learned through the video content.

Assessments of parent and child symptoms will occur at pre-test before LightBEAM begins (T1), immediately after the last week of the LightBEAM intervention (post-test, T2), and 6-month follow-up (T3).

The LightBEAM program offers a promising solution to addressing elevated parental mental health symptoms, parenting stress, and related metrics of child well-being. By adapting BEAM, an evidence-based parenting and mental health app, into LightBEAM, a large-scale online intervention, the present trial aims to provide accessible mental health support for Canadian families. LightBEAM could reach families in remote areas with limited services, offer interim support during waitlists, or function as a self-referral program.

DETAILED DESCRIPTION:
Early childhood is a formative period in which the parent-child relationship plays a central role in child cognitive and social development. When parents of young children experience elevated distress (e.g., depression, anxiety, and anger), it can disrupt healthy parent-child relationships, putting children at risk for negative outcomes, including difficult temperaments, altered cognitive development, and socioemotional risks. Parental distress also can increase children's stress levels, heightening their risk for mental health challenges through both genetic and environmental pathways. The severity of parental distress has been linked to worse child developmental outcomes, but research shows that improving parental mental health can positively impact child functioning. Providing parents with effective mental health support can mitigate the adverse effects of parental distress on children and interrupt the cycle of mental health challenges within families. However, despite the significant impact of untreated parental distress on child development, families face numerous obstacles to accessing timely and effective mental health resources. Some barriers include long wait times and limited availability of affordable services. These barriers increase the risk of cognitive and socioemotional challenges for children.

In response to this growing need, the BEAM (Building Emotional Awareness and Mental Health) program was launched as an app-based intervention that integrates parenting and mental health supports for parents. BEAM offers expert-led videos and activities, online group forums, progress monitoring, and facilitated support through telehealth sessions with parent-peer coaches. The program has demonstrated success in reducing parental anxiety, anger, and sleep difficulties, as well as in improving parent-child interactions. Building on BEAM's success, the investigators translated BEAM into LightBEAM, a massive online open intervention designed to deliver accessible mental health support through an app-based platform. The LightBEAM program is designed with four key components to provide comprehensive support for parenting and mental health: (1) weekly parenting and mental health videos, (2) weekly progress tracking, (3) a group forum, and (4) weekly exercises/activities. Each week, participants will have access to professionally produced psychoeducational videos that offer evidence-based information on topics such as managing stress, fostering positive parent-child interactions, and promoting emotional well-being. Alongside the videos, participants will complete weekly progress tracking to monitor changes in their emotional health and parenting experiences, helping them identify patterns and track their progress over time. To foster a sense of community, the program also features a moderated group forum where parents can connect, share experiences, and provide mutual support. Additionally, participants will engage in weekly exercises designed to reinforce the skills and strategies introduced in the videos. Parent participants have the option to invite a co-parent or other primary caregiver to participate in the LightBEAM program alongside them.

Massive online open interventions, such as LightBEAM, provide evidence-based behavioural support via websites or apps, and allow participants to engage autonomously. This format increases scalability by removing barriers associated with traditional services, such as limited clinician availability and high costs. However, massive online interventions are not without limitations. They may lack the direct clinical oversight needed for individuals requiring more personalized support. While such interventions hold promise for broad mental health service delivery, further research is necessary to evaluate their effectiveness. Thus, this trial will assess the effectiveness and potential of the LightBEAM program through three primary objectives. First, it will evaluate the feasibility and acceptability of the program by examining recruitment and retention rates, participant satisfaction, and the identification of unmet needs. Second, the trial will measure the efficacy of LightBEAM in improving family outcomes by comparing it to a waitlist control group. Key outcomes for parents include emotional well-being and parenting quality, while outcomes for children focus on well-being and socioemotional development. Finally, the trial will identify subgroups of participants who demonstrate the greatest engagement and improvement, using this information to promote equity and inform future program development.

By translating BEAM into LightBEAM, the investigators aim to create a scalable mental health program for families. LightBEAM has the potential to serve families in remote areas with limited access to in-person services, provide interim support during waitlists for individualized care, and function as a self-referral program. By addressing parental mental health, LightBEAM may improve family dynamics and child development, helping to mitigate the negative effects of parental distress.

ELIGIBILITY:
Inclusion Criteria:

* identify as a primary caregiver of any gender to an 18- to 107-month-old child
* reside in Canada with access to internet connection
* be aged 18 years or older
* able to understand/read/speak in English
* report at least mild emotional distress across depression, anxiety, anger, or parenting stress symptoms as assessed by the PHQ-9, GAD-7, PROMIS-Anger, and PSI
* have access to an electronic device

Exclusion Criteria:

* below the age of 18 years
* parenting a child outside the designated age range
* live outside Canada
* have participated in previous iterations of BEAM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in parent mental health symptom composite. | All measures to be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  The parent mental health composite score will be defined uniquely for each participant using a weighted average of their pre-intervention (T1) mental health profile (i.e., self-report symptoms of depression, anxiety, anger, sleep problems, and parenting stress). Pre-intervention symptoms above established clinical cut-offs will be mean-centred, standardized, and included in the participant's composite mental health symptom score weighted by the symptom's pre-intervention severity. In this way, the primary outcome will track mean change in each participant's most clinically elevated pre-intervention symptoms.
  This composite will use validated measures of depression symptom severity (Patient Health Questionnaire-9), anxiety symptom severity (Generalized Anxiety Disorder-7), anger (PROMIS Anger), sleep disturbances (PROMIS Sleep Disturbance), and parenting stress (Parenting Stress Index - 4th Edition - Short Form). Change in each measure is also a secondary outcome, described below.
Feasibility and Acceptability of LightBEAM program. | To be assessed pre-intervention (T1), during intervention, and immediately after intervention (T2).
  Acceptability and uptake of the LightBEAM program will be assessed in three ways: (1) rates of attrition, (2) qualitative analysis of responses to post-intervention focus group questions that probe barriers and facilitators to program engagement, and (3) program engagement measures from back-end app data (e.g., number of logins, time spent on the app, forum posts, number of videos watched).

SECONDARY OUTCOMES:
Change in parent depressive symptoms. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Parent depressive symptoms will be measured using the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a self-report measure of depression symptom severity. Total scores range from 0 to 27, with higher scores indicating more severe depression symptoms.
Change in parent anxiety symptoms. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Parent anxiety symptoms will be measured using the Generalized Anxiety Disorder questionnaire (GAD-7). The GAD-7 is a self-report measure of anxiety symptom severity. Total scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Change in parent anger symptoms. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Parent anger symptoms will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Anger scale. The PROMIS-Anger is a self-report measure of anger symptoms. Total scores range from 5 to 25, with higher scores indicating more anger symptoms.
Change in parent self-compassion. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Parent self-compassion will be measured using the Self-Compassion Scale Short Form (SCS-SF) Questionnaire. The SCS-SF is a self-report measure of self-compassion. Scores range from 12 to 60, and a mean score is computed. Means lay between 1 and 5, with higher mean scores indicating higher levels of self-compassion.
Changes in parent sleep problems. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Parent sleep problems will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance scale. The PROMIS-Sleep Disturbance is a self-report measure of sleep disturbances. Total scores range from 8 to 40, with higher scores indicating more severe sleep disturbances.
Change in parenting stress. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Parenting stress will be measured using the Parenting Stress Index - 4th Edition - Short Form (PSI-4-SF). The PSI-4-SF is a self-report measure that captures three sources of stress; from parent stress, from a difficult child, and from parent-child interactions. Total scores range from 36 to 180, with higher scores indicating more parenting stress.
Change in harsh parenting disciplinary practices. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Harsh parenting practices will be measured using 10 items measuring Overreactivity from The Parenting Scale (PS-Overreactivity). The PS-Overreactivity is a self-report measure of parenting behavior and dysfunctional discipline in parents with young children. Total scores range from 10 to 70, with higher scores indicating higher levels of ineffective discipline practices.
Change in child behaviour. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Child behaviour will be measured using the Child Behaviour Checklist (CBCL). The CBCL is a parent-report measure of emotional and behavioural problems in children. Total scores range from 0 to 198, with higher scores indicating more emotional and behavioural challenges.
Change in co-parent mental health symptom composite. | All measures to be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  The co-parent mental health composite score will be defined uniquely for each participant using a weighted average of their pre-intervention (T1) mental health profile (i.e., self-report symptoms of depression, anxiety, anger, sleep problems, and parenting stress). Pre-intervention symptoms above established clinical cut-offs will be mean-centred, standardized, and included in the participant's composite mental health symptom score weighted by the symptom's pre-intervention severity. In this way, the primary outcome will track mean change in each participant's most clinically elevated pre-intervention symptoms.
  This composite will use validated measures of depression symptom severity (Patient Health Questionnaire-9), anxiety symptom severity (Generalized Anxiety Disorder-7), anger (PROMIS Anger), sleep disturbances (PROMIS Sleep Disturbance), and parenting stress (Parenting Stress Index - 4th Edition - Short Form). Change in each measure is also a secondary outcome.
Change in co-parent depressive symptoms. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Co-parent depressive symptoms will be measured using the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a self-report measure of depression symptom severity. Total scores range from 0 to 27, with higher scores indicating more severe depression symptoms.
Change in co-parent anxiety symptoms. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Co-parent anxiety symptoms will be measured using the Generalized Anxiety Disorder questionnaire (GAD-7). The GAD-7 is a self-report measure of anxiety symptom severity. Total scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Change in co-parent anger symptoms. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Co-parent anger symptoms will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Anger scale. The PROMIS-Anger is a self-report measure of anger symptoms. Total scores range from 5 to 25, with higher scores indicating more anger symptoms.
Change in co-parent self-compassion. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Co-parent self-compassion will be measured using the Self-Compassion Scale Short Form (SCS-SF) Questionnaire. The SCS-SF is a self-report measure of self-compassion. Scores range from 12 to 60, and a mean score is computed. Means lay between 1 and 5, with higher mean scores indicating higher levels of self-compassion.
Changes in co-parent sleep problems. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Co-parent sleep problems will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance scale. The PROMIS-Sleep Disturbance is a self-report measure of sleep disturbances. Total scores range from 8 to 40, with higher scores indicating more severe sleep disturbances.
Change in co-parent parenting stress. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Co-parent parenting stress will be measured using the Parenting Stress Index - 4th Edition - Short Form (PSI-4-SF). The PSI-4-SF is a self-report measure that captures three sources of stress; from parent stress, from a difficult child, and from parent-child interactions. Total scores range from 36 to 180, with higher scores indicating more parenting stress.
Change in co-parent harsh parenting disciplinary practices. | To be assessed pre-intervention (T1), immediately after intervention (T2), at 6-month follow-up (T3).
  Harsh parenting practices in co-parents will be measured using 10 items measuring Overreactivity from The Parenting Scale (PS-Overreactivity). The PS-Overreactivity is a self-report measure of parenting behavior and dysfunctional discipline in parents with young children. Total scores range from 10 to 70, with higher scores indicating higher levels of ineffective discipline practices.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
Summary statistics (e.g., questionnaire subscales, sociodemographics, aggregated forum usage data) paired with non-identifiable participant IDs may be shared on data repositories such as the Open Science Framework.

REFERENCES:
- [Background] Muñoz, R. F., Bunge, E. L., Chen, K., Schueller, S. M., Bravin, J. I., Shaughnessy, E. A., & Pérez-Stable, E. J. (2016). Massive open online interventions: A novel model for delivering behavioral-health services worldwide. Clinical Psychological Science, 4(2), 194-205. https://doi.org/10.1177/2167702615601185
- [Background] Letourneau NL, Dennis CL, Benzies K, Duffett-Leger L, Stewart M, Tryphonopoulos PD, Este D, Watson W. Postpartum depression is a family affair: addressing the impact on mothers, fathers, and children. Issues Ment Health Nurs. 2012 Jul;33(7):445-57. doi: 10.3109/01612840.2012.673054. PMID 22757597
- [Background] Keller PS, Kouros CD, Erath SA, Dahl RE, El-Sheikh M. Longitudinal relations between maternal depressive symptoms and child sleep problems: the role of parasympathetic nervous system reactivity. J Child Psychol Psychiatry. 2014;55(2):172-9. doi: 10.1111/jcpp.12151. Epub 2013 Oct 9. PMID 24117807
- [Background] Hammen, C. (2002). Context of stress in families of children with depressed parents. In Children of depressed parents: Mechanisms of risk and implications for treatment (pp. 175-199). American Psychological Association. https://doi.org/10.1037/10449-007
- [Background] Giannakopoulos G, Solantaus T, Tzavara C, Kolaitis G. Mental health promotion and prevention interventions in families with parental depression: A randomized controlled trial. J Affect Disord. 2021 Jan 1;278:114-121. doi: 10.1016/j.jad.2020.09.070. Epub 2020 Sep 15. PMID 32956960
- [Background] Joyce KM, Rioux C, MacKinnon AL, Katz LY, Reynolds K, Kelly LE, Klassen T, Afifi TO, Mushquash AR, Clement FM, Chartier M, Xie EB, Penner KE, Hunter S, Berard L, Tomfohr-Madsen L, Roos LE. The Building Emotional Awareness and Mental health (BEAM) program developed with a community partner for mothers of infants: protocol for a feasibility randomized controlled trial. Pilot Feasibility Stud. 2023 Mar 9;9(1):35. doi: 10.1186/s40814-023-01260-y. PMID 36895006
- [Background] Xie EB, Simpson KM, Reynolds KA, Giuliano RJ, Protudjer JLP, Soderstrom M, Sauer-Zavala S, Giesbrecht GF, Lebel C, Mackinnon AL, Rioux C, Penner-Goeke L, Freeman M, Salisbury MR, Tomfohr-Madsen L, Roos LE. Building Emotional Awareness and Mental Health (BEAM): study protocol for a phase III randomized controlled trial of the BEAM app-based program for mothers of children 18-36 months. Trials. 2022 Sep 5;23(1):741. doi: 10.1186/s13063-022-06512-5. PMID 36064436
- [Background] MacKinnon AL, Simpson KM, Salisbury MR, Bobula J, Penner-Goeke L, Berard L, Rioux C, Giesbrecht GF, Giuliano R, Lebel C, Protudjer JLP, Reynolds K, Sauer-Zavala S, Soderstrom M, Tomfohr-Madsen LM, Roos LE. Building Emotional Awareness and Mental Health (BEAM): A Pilot Randomized Controlled Trial of an App-Based Program for Mothers of Toddlers. Front Psychiatry. 2022 Jun 24;13:880972. doi: 10.3389/fpsyt.2022.880972. eCollection 2022. PMID 35815022
- See also: LightBEAM Program Website — https://www.thelightbeamprogram.com/